CLINICAL TRIAL: NCT02525484
Title: A Phase I, Open-Label, Randomized, Four-Treatment Period, Four-Sequence, Single-Dose, Crossover, Pharmacokinetic Bioequivalence Study Comparing Pirfenidone Tablet and Capsule Dosage Forms in Healthy Adult Volunteers
Brief Title: A Bioequivalence Study Comparing Pirfenidone Tablet and Capsule Dosage Forms in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GP29830
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — pirfenidone

ARMS (4):
- Pirfenidone ACBD treatment sequence (Experimental): Participants will be given 801 milligrams (mg) single oral doses of pirfenidone on Days 1, 4, 7 and 10 during the study. Participants will be administered, capsules (3 x 267-mg capsule) in fed state (treatment A) on Day 1 and in fasted state (treatment C) on Day 4, 801-mg tablet in fed state (treatment B) on Day 7 and in fasted state (treatment D) on Day 10.
  Interventions: Drug: Pirfenidone
- Pirfenidone BADC treatment sequence (Experimental): Participants will be given 801 mg single oral doses of pirfenidone on Days 1, 4, 7 and 10 during the study. Participants will be administered, 801-mg tablet in fed state (treatment B) on Day 1, capsules (3 x 267-mg capsule) in fed state (treatment A) on Day 4, 801-mg tablet in fasted state (treatment D) on Day 7 and capsules (3 x 267-mg capsule) in fasted state (treatment C) on Day 10.
  Interventions: Drug: Pirfenidone
- Pirfenidone CDAB treatment sequence (Experimental): Participants will be given 801 mg single oral doses of pirfenidone on Days 1, 4, 7 and 10 during the study. Participants will be administered, capsules (3 x 267-mg capsule) in fasted state (treatment C) on Day 1, 801-mg tablet in fasted state (treatment D) on Day 4, capsules (3 x 267-mg capsule) in fed state (treatment A) on Day 7 and 801-mg tablet in fed state (treatment B) on Day 10.
  Interventions: Drug: Pirfenidone
- Pirfenidone DBCA treatment sequence (Experimental): Participants will be given 801 mg single oral doses of pirfenidone on Days 1, 4, 7 and 10 during the study. Participants will be administered, 801-mg tablet in fasted state (treatment D) on Day 1 and in fed state (treatment C) on Day 4, capsules (3 x 267-mg capsule) in fasted state (treatment C) on Day 7 and in fed state (treatment A) on Day 10.
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone 801 mg single oral doses will be given either in the form of tablet or capsules under fed or fasted conditions on Days 1, 4, 7 and 10.

SUMMARY:
This is a Phase I, open-label, randomized, four-treatment period, four-sequence, single-dose, crossover pharmacokinetic study to determine the bioequivalence of pirfenidone after administration of tablet and capsule dosage forms under both fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 55 years of age, inclusive, at the time of screening
* Participants of body mass index of 18.5-30.0 kilograms per square meter (kg/m^2), inclusive
* Participants of reproductive potential must be willing to use reliable contraceptive methods

Exclusion Criteria:

* Participants with significant medical history or unstable hepatic, pulmonary, metabolic, neurologic, cardiovascular, gastrointestinal, hematologic, or psychiatric systems, in the opinion of the investigator that may alter the absorption, metabolism, or elimination of study drug
* Participants with calculated creatinine clearance rate less than (<) 30 milliliters per minute (mL/min) (calculated using the Cockcroft-Gault equation) at screening
* Participants with any use of, or intent to use, medications, including prescription, over-the-counter, herbal preparations, or vitamin/mineral supplementation other than study medications from 14 days before screening through the follow-up telephone call (except for contraception purpose)
* Participants who have received fluvoxamine therapy within 28 days before screening
* Participants who have received any medications known to chronically alter drug absorption, metabolism, or elimination processes within 28 days of screening, or participants who are taking drugs known to affect liver function, in the opinion of the Sponsor or investigator
* Participants who have taken investigative drug and/or device in another clinical study within 28 days or within the investigational drug 5 half-lives, whichever is longer, before screening
* Participants previously dosed in any pirfenidone clinical study
* Participants with any hypersensitivity or idiosyncratic reaction to pirfenidone or the constituents of pirfenidone
* Participants with any elevation of liver test results (alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase [GGT], direct bilirubin, or alkaline phosphatase above the upper limit of normal)
* Participants with the following hemoglobin levels at screening: males < 13.5 grams per deciliter (g/dL), females < 11.5 g/dL
* Females with a positive serum pregnancy test or who are breastfeeding
* Participants who are seropositive for hepatitis B surface antigen, hepatitis C virus antibodies, or human immunodeficiency (HIV) antibodies at screening
* Participants who have a clinically significant abnormal electrocardiogram (ECG) at screening or a Fridericia corrected QT interval (QTcF) greater than (>) 500 milliseconds (ms) at screening
* Participants with a plasma donation within 28 days before screening or with a donation of blood or blood products or significant blood loss within 56 days before screening
* Participants with poor venous access
* Participants who have used cigarettes (including vapor cigarettes), cigars, and nicotine-containing products within 3 months before screening or plan to use them through completion of the follow-up telephone call
* Participants with a history of alcoholism or drug abuse, per discretion of the investigator, within 2 years of screening or a positive qualitative drug screen for drugs of abuse at screening or Day -1
* Participants who have not withheld alcoholic beverages/alcohol-containing products or caffeinated beverages/caffeine- or xanthine-containing products at least 72 hours before first study dose administration or who plan to consume them during the study or a positive qualitative drug screen for alcohol at screening or Day -1
* Participants with an abnormal diet (as determined by the investigator) within the 28 days before first study dose administration
* Participants who have not withheld consuming cruciferous vegetables (broccoli, kale, Brussels sprouts), grapefruit or grapefruit juice, or chargrilled meat 48 hours before dosing or who plan to consume them during the study
* Participants who cannot refrain from strenuous exercise from 48 hours before first study dose administration through completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Pirfenidone | 11 days
Area Under the Plasma Concentration Versus Time Curve (AUC) from Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-t]) of Pirfenidone | 11 days
AUC from Time Zero to Infinity (AUC[0-inf]) of Pirfenidone | 11 days

SECONDARY OUTCOMES:
Ratio of AUC(0-t) to AUC(0-inf) of Pirfenidone | 11 days
Terminal Elimination Rate Constant of Pirfenidone | 11 days
Apparent Terminal Half-Life (t1/2) of Pirfenidone | 11 days
Time to Peak Plasma Concentration of Pirfenidone | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Merritt Island, Florida, United States